CLINICAL TRIAL: NCT03815903
Title: A Phase 3, Randomized, Open-label Clinical Trial of Induction Chemotherapy Followed by Chemoradiotherapy Versus Chemoradiotherapy in Patients With Locally Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: Induction Chemotherapy for Locally Advanced Head and Neck Squamous Cell Carcinoma
Acronym: INDUCTION
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Barretos Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BarretoCH - 201801
Record Dates: First submitted 2018-12-19; First posted 2019-01-24 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2018-12

CONDITIONS: Locally Advanced Malignant Neoplasm
MeSH Terms: interventions — Induction Chemotherapy; Chemoradiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A - induction chemotherapy (Active Comparator)
  Interventions: Drug: Induction chemotherapy; Combination Product: Chemoradiotherapy
- B - chemoradiotherapy (Experimental)
  Interventions: Combination Product: Chemoradiotherapy

INTERVENTIONS:
Drug: Induction chemotherapy — 3 cycles, each 21 days, of Cisplatin 80mg/m2 plus Paclitaxel 175mg/m2
  Arms: A - induction chemotherapy
Combination Product: Chemoradiotherapy — Radiotherapy 70Gy convencional fractionation concomitant to 3 cycles, each 21 days, of Cisplatin 100mg/m2

SUMMARY:
The benefit of induction chemotherapy followed by chemoradiotherapy for locally advanced head and neck squamous cell carcinoma is unknown. The present study is investigating if this therapeutic strategy improve overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed histological diagnosis of squamous cell carcinoma or undifferentiated carcinoma of the oropharynx, hypopharynx or larynx;
* Locally advanced stage (stage IVa / b - AJCC 8th edition), classified as resectable ** or unresectable and candidate for treatment based on radiotherapy and chemotherapy;
* Locally advanced stage (stage III - AJCC 8th edition), classified as resectable or unresectable, positive p16 and candidate for treatment based on radiotherapy and chemotherapy;
* It will be allowed to include a patient with cervical lymphadenectomy if the primary lesion is measurable;
* Presence of measurable disease according to RECIST 1.1 criteria;
* ECOG performance status of 0-1;
* ≥ 18 years;
* Adequate marrow reserve indicated by:

  * Absolute neutrophil count (ANC) ≥ 1500 / mm³ or Platelets> 100,000 / mm³
  * Hemoglobin ≥ 9 g / dL - red blood cell transfusion will be allowed in the screening period if necessary
* Adequate renal and hepatic function:

  * Serum bilirubin ≤ 1.5 times the upper limit of normal the TGO and TGP ≤ 3 upper limit of normal. If hepatic metastasis ≤ 5 upper limit of normal
  * Serum creatinine ≤ 1.5 mg / dL and creatinine clearance ≥ 60 mL / min calculated by Cockcroft-Gault.

Exclusion Criteria:

* Patient submitted to curative resection of the primary site and / or metastatic site. NOTE: Patients submitted to cervical lymphadenectomy without surgery to the primary tumor are eligible;
* Radiation therapy or previous chemotherapy for head / neck tumor;
* Patients with occult primary tumor;
* T4 from any site, resectable, with invasion of cartilage or jaw;
* History of BMT or stem cell therapy;
* Synchronous tumor or previous history of neoplasia, except for in situ carcinoma of the cervix, basal cell carcinoma or epidermoid carcinoma. Patients with previous history of cancer already treated and without evidence of disease for more than 3 years may participate in the study;
* Prophylactic use of G-CSF or GM-CSF two weeks prior to the study;
* Clinically significant heart disease: unstable angina or myocardial infarction 6 months prior to study entry Symptomatic ventricular arrhythmia the ICC classified as NYHA ≥ II • Uncontrolled hypercalcemia;
* Uncontrolled infection;
* Any other comorbidity that the investigator's judgment is inappropriate for the study;
* Peripheral neuropathy> grade 2;
* Hearing loss> grade 2;
* Known positive serology for hepatitis B, hepatitis C or HIV
* Use of antiretrovirals;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 434 (Estimated)
Dates: Start 2018-12-19 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
3-years overall survival | From date of randomization until 3 years

SECONDARY OUTCOMES:
Progression free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  PFS
Systemic relapse free survival | From date of randomization until the date of first systemic relapse or date of death from any cause, whichever came first, assessed up to 100 months
Overall survival | From date of randomization until the date of death from any cause, whichever came first, assessed up to 100 months
Overall response rate | At the end of Cycle 3 of IC (each cycle is 21 days) and 8 weeks after the end of radiotherapy, through study completion, an average of 6 months
Adverse Events Rates | At the end of cycle 1, cycle 2 and cycle 3 (each cycle is 21 days).
1-year functional organ preservation rate | From date of randomization until 1 year after
Quality of Life (EORTC Quality of Life Questionnare - C30 version 3.0) | From date of randomization until 5 years
  The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Overall response rate to induction chemotherapy | At the end of Cycle 3 (each cycle is 21 days)

CONTACTS AND LOCATIONS:
Locations (1):
- Barretos Cancer Hospital, Barretos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided